CLINICAL TRIAL: NCT01572181
Title: Phase 2 Study of a Reduced-toxicity Myeloablative Conditionning Regimen Using Fludarabine and Full Doses of iv Busulfan in Pediatric Patients Not Eligible for Standard Myeloablative Conditioning Regimens
Brief Title: Study of a Reduced-toxicity Myeloablative Conditioning Regimen Using Fludarabine and Full Doses of Intravenous Busulfan in Pediatric Patients Not Eligible for Standard Myeloablative Conditioning Regimens
Acronym: FB4-PEDIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/11/06-N
Record Dates: First submitted 2012-02-21; First posted 2012-04-06 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Busulfan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drugs (Experimental): Fludarabine IV- Busulfan IV (Busilvex®) - Anti-thymocyte globulines (Thymoglobuline®)
  Interventions: Drug: Fludarabine IV- Busulfan IV (Busilvex®) - Anti-thymocyte globulines (Thymoglobuline®)

INTERVENTIONS:
Drug: Fludarabine IV- Busulfan IV (Busilvex®) - Anti-thymocyte globulines (Thymoglobuline®) — * IV fludarabine (30 mg/m²/day for 5 days)
  * IV Busulfan (Busilvex 3.2 mg/kg/day for 4 days) (the Busulfan dose is to be adapted to the weight of the child according to the drug label)
  * Anti-thymocyte globulines (Thymogolubuline, 2.5 mg/kg/day for 2 days).

SUMMARY:
The purpose of this study is to assess transplant-related mortality (TRM) at one year after allogeneic hematopoietic stem cell transplantation (allo-HSCT) prepared by a "reduced toxicity myeloablative" conditioning regimen in young patients (children and adolescents) with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria

* Children and adolescents aged over 12 months and under 25 years
* Availability of an HLA identical family donor or an HLA-matched unrelated donor (10/10 or 9/10 if the mismatch level is at HLACw for an unrelated donor) or availability of an HLA matched cord blood (5/6 or 6/6)
* Informed consent signed by patients (18-25 years) and patient's legal representative, parent(s) or guardian (cf p13)
* Diagnosis of a hematologic malignancy which is a candidate for allo-HSCT, but not eligible for standard or conventional myeloablative conditioning regimens because of high risk for toxicity.
* Are considered as criteria of non-eligibility for standard or conventional myeloablative conditioning:

  * a history of autologous or allogeneic stem cell transplantation
  * comorbidities or medical history predictive of a prohibitive rate of TRM and toxicity with the use of standard high dose chemotherapy and / or radiotherapy.

Exclusion Criteria:

* Patient has been administered any other systemic chemotherapeutic drug (including Gemtuzumab) within 21 days prior to trial enrollment and start of the conditioning regimen. Hydroxyurea is permitted if indicated to control induction refractory disease, and IT chemotherapy is allowed if indicated as maintenance treatment for previously diagnosed leptomeningeal disease, that has been in remission for at least 3 months prior to enrollment on this study.
* Active infection. Protocol PI will be final arbiter if there is uncertainty regarding whether a previous infection is resolved.
* Children and adolescents who are not older than 12 months and under 25 years
* A donor who is HLA mismatched at the level of more than one locus.
* Poor performance status (Lansky < 50%)
* Life expectancy is severely limited by concomitant illness and expected to be <12 weeks.
* Left ventricular ejection fraction < 30%. Uncontrolled arrhythmias or symptomatic cardiac disease.
* Symptomatic pulmonary disease. FEV1, FVC and DLCO <30% of expected corrected for hemoglobin.
* Creatinine clearance less than 30 mL/m per 1.73 m2 or requiring dialysis
* Evidence of chronic active hepatitis or cirrhosis. If positive hepatitis serology, discuss with Study Chairman and consider liver biopsy.
* Effusion or ascites >1L prior to drainage.
* HIV-positive.
* Female pregnancy
* Absence of effective contraception among boys and girls of childbearing potential (that contraception should be continued until 6 months after stopping treatment)
* Breastfeeding
* Patient's legal representative, parent(s) or guardian not able to sign informed consent.
* children's refusal
* Hypersensitivity to rabbit proteins, to the active substance or to any of the excipients of experimental products

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Transplant-related mortality (TRM) | 12 months
  Evaluation of the cumulative incidence of TRM at 12 months after transplantation

SECONDARY OUTCOMES:
Incidence of engraftment | Day+42
  Incidence of engraftment defined as the first day of neutrophil (>500/μl for 3 consecutive days). Engraftment failure is defined as neutrophil <500/μl at day+42 after allo-SCT.
Evaluation of overall (OS) and disease-free survival (DFS) | 12 months
  Evaluation of overall (OS) and disease-free survival (DFS) at 1 year after transplantation
Cumulative incidence of relapse, death from disease, and non-relapse mortality (NRM) | 12 months
  Cumulative incidence of relapse, death from disease, and non-relapse mortality (NRM)
Cumulative incidences and severity of acute and chronic Graft-versus-Host disease | 12 months
  Cumulative incidences and severity of acute and chronic Graft-versus-Host disease
Immune Recovery (to be determined in a subgroup of patients) | 12 months
  Immune Recovery parameters: blood counts, bone marrow aspiration with evaluation of morphological response.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, Professor, Principal Investigator — Nantes University Hospital
Locations (15):
- France (15):
  - University Hospital, Besançon
  - University Hospital, Bordeaux
  - University Hospital, Clermont-Ferrand
  - University Hospital, Grenoble
  - University Hospital, Lille
  - University Hospital, Lyon
  - University Hospital, Marseille
  - University Hospital, Montpellier
  - University Hospital, Nancy
  - University Hospital, Nantes
  - University Hopsital, Paris
  - University Hospital, Paris
  - University Hospital, Rennes
  - University Hopsital, Rouen
  - University Hospital, Strasbourg

REFERENCES:
- [Derived] Rialland F, Grain A, Labopin M, Michel G, Gandemer V, Paillard C, Pochon C, Clement L, Brissot E, Jubert C, Sirvent A, Rohrlich PS, Plantaz D, Dalle JH, Mohty M. Reduced-toxicity myeloablative conditioning regimen using fludarabine and full doses of intravenous busulfan in pediatric patients not eligible for standard myeloablative conditioning regimens: Results of a multicenter prospective phase 2 trial. Bone Marrow Transplant. 2022 Nov;57(11):1698-1703. doi: 10.1038/s41409-022-01769-5. Epub 2022 Aug 26. PMID 36028757